CLINICAL TRIAL: NCT04880538
Title: Enteric Neural Precursor Cells (ENPC) in the Human Gut - Identification of Molecular Signature and Characterization of Their Proliferative & Neurogenic Potential Using Surgical/Endoscopic Biopsies in Vitro
Brief Title: Enteric Neural Precursor Cells (ENPC) in the Human Gut
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00146589
Record Dates: First submitted 2021-04-30; First posted 2021-05-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Gastrointestinal Dysmotility
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endoscopic GI tract biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Asymptomatic patients for any motility disorder: Asymptomatic patients for any motility disorder
  Interventions: Procedure: Endoscopic procedure
- Patients with gastrointestinal dysmotility: Patients with gastrointestinal dysmotility
  Interventions: Procedure: Endoscopic procedure

INTERVENTIONS:
Procedure: Endoscopic procedure — Endoscopic biopsy of one or more of the following: esophagus, stomach, small bowel, colon, or rectum as part of patient clinical care. Biopsies will be performed during endoscopy or colonoscopy and will be transported to the research laboratory for evaluation.

SUMMARY:
The study aim is to acquire human tissues to (a) understand the structure and organization of the human Enteric Nervous System; (b) perform a molecular transcriptomic profile of individual cells residing in the human gut; (c) study the turnover rates of individual cell types by Fluorescence-activated cell sorting-aided C14 dating of cells; and finally (d) culture the human gut-derived cells characterize the human adult enteric neural stem cell and study its potential for Neuro-glial differentiation. This study will advance our knowledge of the the cellular and molecular correlates of changes in the Enteric Nervous System that are associated with disorders of motility.

DETAILED DESCRIPTION:
(i) To study the structure and organization of the human Enteric Nervous System by tissue clarification, immunofluorescence, and 2-photon and light-sheet microscopy.

(ii) To find out the molecular signature that defines various gastrointestinal cells that include the neurons, glia, precursor cells within the Enteric Nervous System and cells associated with the Enteric Nervous System, such as Interstitial Cell of Cajal and macrophages in the human whole gut surgical resection and full thickness endoscopic resection-derived tissues using single cell RNA sequencing and analyses.

(iii) To isolate these cells and study their proliferative and neurogenic potential in vitro and on transplantation into the gut tissue of immunodeficient mice.

(iv) To time stamp and determine the age of Enteric Nervous System cells in adults and determine whether different enteric disease states alter the cycling times of these cells.

(v) To use gut specimens derived from surgical resections and full thickness endoscopic resection-derived tissues for

1. Generating ex vivo preps to study and understand the electrophysiological properties of the gut wall and
2. Generating cultured ex vivo preps to understand the interaction between enteric extracellular matrix and cells of the Enteric Nervous System.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patients in the age range 18 - 100.
* Patients suffering from Irritable Bowel Syndrome, Inflammatory Bowel Disease, Diabetes, Gastroparesis, will be included.
* Patients suffering from Collagen disorders such as Alport Syndrome, Ehlers-Danlos Syndrome, Goodpasture Syndrome.
* Patients suffering from plexiform neurofibromas.
* Patients with bariatric surgery.
* Patients with appendicitis.
* Patients with scleroderma.

Exclusion Criteria:

* Patients suffering from HIV, Hepatitis C, and other infectious diseases that require the handling of tissues in a Bio-safety level 3 environment.
* Patients suffering from infectious enteric disorders.
* Patients without any Gastrointestinal disorders (i.e. healthy volunteers).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal diseases.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Visualization of the network of Nestin+ cells in human gut resection specimens. | Up to one year
  Presence or absence of antibodies (including but not limited to) specific to Nestin, p75 neurotrophin receptor, pan-neuronal antibodies, pan-glial antibodies, antibodies against Interstitial Cells of Cajal.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Hui, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States